CLINICAL TRIAL: NCT03583034
Title: Prospective Assessment of Outcomes and Complications of Patients Submitted to Holmium Laser Enucleation of the Prostate (HoLEP) in a High Volume Center
Brief Title: Outcomes and Complications of Holmium Laser Enucleation of the Prostate in Expert Hands
Acronym: ExpHo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Francesco Montorsi, Chairman Department of Urology IRCCS San Raffaele Hospital Professor of Urology Vita Salute San Raffaele University, IRCCS San Raffaele
Other Study IDs: ExpHo study
Record Dates: First submitted 2018-06-18; First posted 2018-07-11 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: HoLEP; Prostate
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Holmium laser enucleation of the prostate (HoLEP) — Surgery for benign prostatic hyperplasia

SUMMARY:
The efficacy and safety of holmium laser enucleation of the prostate (HoLEP) for the treatment of lower urinary tract symptoms (LUTS) associated with benign prostatic hyperplasia (BPH) have been comprehensively assessed. However, HoLEP is considered as a challenging procedure with a steep learning curve. As such, HoLEP is not as yet considered the gold standard for the surgical treatment of LUTS/BPH by international clinical guidelines.

The investigators aim to assess the complications and outcomes of patients treated with HoLEP by high volume surgeons, in order to provide data on the safety of the procedure and identify the profile of patients who may benefit from a dedicated clinical management to reduce the risk of post-operative complications.

DETAILED DESCRIPTION:
This is a prospective case-series study collecting data of patients treated with HoLEP at a single academic center. Patients submitted to surgery for bladder outlet obstruction (BOO) due to BPH will be consecutively included. All surgeries will be performed by two experienced surgeons with more than 1000 procedures performed (FM; GB).

Patients with neurological diseases and those with a history of previous surgery of the lower urinary tract (e.g. urethra and prostate surgery) will be excluded.

At the time of primary screening, all patients will be assessed with a comprehensive medical history; other pre-operative data will include: prostate volume (as assessed with trans-rectal prostate ultrasound); uroflowmetry parameters; total Prostate specific Antigen (PSA); baseline haemoglobin and creatinine level. Moreover, all patients will be invited to fill psychometric validated questionnaires assessing pre-operative urinary and sexual function, thus including: the International Prostatic Symptoms Score (IPSS); the International Index of Erectile Function (IIEF); the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF); and the Overactive Bladder Questionnaire (OABq). Moreover, urinary continence (UC) will be further assessed with a single question, and UC defined as no-pad use. Patients' medications will be also recorded.

Intra-operative data will be collected at the time of surgery, including: patients' systolic blood pressure; laser settings; enucleation efficiency (weight of enucleated tissue divided by lasing time) and morcellation efficiency (weight of enucleated tissue divided by morcellation time). Moreover, surgeons will be requested to provide a subjective estimation of the difficulty of the procedure with a 10-point Likert scale.

Post-operative data including: length of stay; timing of catheter removal and complications, will be also collected.

All patients will be re-assessed at 1 week after surgery to check for UC. Subjective symptoms, as assessed with validated questionnaires (IPSS; IIEF, ICIQ-SF; OABq), along with post-operative complications and medications used, will be firstly assessed at 1 month after surgery. All patients will undergo a first uroflowmetry evaluation at 3 months after surgery; at this time-point data on blood tests (total PSA, haemoglobin and creatinine), urine culture and symptoms scores will be collected.

A final assessment will be performed at 1 year after surgery including: blood tests, uroflowmetry, IPSS, IIEF, ICIQ-SF, OABq and complications.

Over the follow-up period, the prevalence of patients needing medications for disturbing symptoms will be recorded; moreover, pelvic floor training (PFT) will be suggested to each patient reporting pad-use for urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lower urinary tract symptoms due to benign prostatic hyperplasia

Exclusion Criteria:

* neurological diseases; previous surgery on the lower urinary tract (urethra/prostate)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients submitted to surgery for bladder outlet obstruction (BOO) due to BPH
Sampling Method: Non-Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-04-18 (Estimated); Study Completion 2020-06-18 (Estimated)

PRIMARY OUTCOMES:
Functional outcomes as assessed with IPSS questionnaire | 12 months
  functional urinary outcomes will be assessed with IPSS questionnaire at different time points over the first year after surgery.

SECONDARY OUTCOMES:
Identification of clinical characteristics associated with risk of post-operative complications (recorded according to the Clavien-Dindo classification) | 12 months
  The association between clinical characteristics (e.g. age, BMI, comorbidities, prostate volume) and the risk of post-operative complications will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, MI, Italy

REFERENCES:
- [Derived] Capogrosso P, Ventimiglia E, Fallara G, Schifano N, Costa A, Candela L, Pellegrino F, Colandrea G, Cignoli D, De Angelis M, Belladelli F, Longoni M, Avesani G, Lanzaro F, Scattoni V, Deho F, Salonia A, Briganti A, Montorsi F. Holmium Laser Enucleation of the Prostate Is Associated with Complications and Sequelae Even in the Hands of an Experienced Surgeon Following Completion of the Learning Curve. Eur Urol Focus. 2023 Sep;9(5):813-821. doi: 10.1016/j.euf.2023.03.018. Epub 2023 Apr 15. PMID 37069007